CLINICAL TRIAL: NCT02052024
Title: Myobloc Atrophy Study
Acronym: MAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Solstice Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USWM-206-1010
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Spasticity Secondary to Either a Disorder or Trauma; Spinal Cord Injury (SCI); Brain Injury; Tumor; Stroke
Keywords: Spasticity; Modified Ashworth Scale; MYOBLOC; Botox; Muscle Atrophy
MeSH Terms: conditions — Wounds and Injuries; Spinal Cord Injuries; Brain Injuries; Neoplasms; Stroke; Muscle Spasticity; Muscular Atrophy | interventions — Botulinum Toxins, Type A; rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Active Comparator): Treatment group will receive 100 units of BOTOX and will receive 1-3 injections per muscle at each visit.
  Interventions: Drug: Botox
- MYOBLOC (Active Comparator): Treatment group will receive 5,000 units of MYOBLOC and will receive 1-3 injections per muscle at each visit.
  Interventions: Drug: MYOBLOC

INTERVENTIONS:
Drug: Botox — Treatment group will receive 100 units of BOTOX and subjects will receive 1-3 injections per muscle at each visit.
  Other Names: Botulinum Toxin Type A
  Arms: Botox
Drug: MYOBLOC — Treatment group will receive 5,000 units of MYOBLOC and subjects will receive 1-3 injections per muscle at each visit.
  Other Names: Botulinum Toxin Type B
  Arms: MYOBLOC

SUMMARY:
The present pilot study is designed to assess the extent to which BOTOX and MYOBLOC cause muscle atrophy in spastic patients. The primary objective is to assess whether there is statistically significant difference in muscle atrophy between the two groups over a one year period.

DETAILED DESCRIPTION:
Botulinum toxin has long been used as a clinical application for the treatment of overactive skeletal and smooth muscles, i.e. spasticity. The benefits of botulinum therapy are indisputable, however, muscle atrophy is one main adverse effect that may hinder a patient's strength and decrease the ability for the practitioner to accurately administer botulinum toxin to a specific muscle group. This, in turn may cause unintentional weakness of adjacent muscle groups through inaccurate targeting or diffusion of botulinum toxin. Currently, only two serotypes (abbreviated to BTX-A (BOTOX, XEOMIN and DYSPORT) and BTX-B (MYOBLOC), respectively) are used in clinical practice for spasticity. Research has shown that both BTX-A and BTX-B are efficacious in the treatment of spasticity. However, there is no documented literature evaluating if there is a statistically significant difference in the degree of muscle atrophy using BTX-A versus BTX-B.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older with spasticity secondary to either a disorder or trauma, such as a spinal cord injury (SCI), a brain injury, a tumor, a stroke, multiple sclerosis (MS), or a peripheral nerve injury.
* Participants must have the ability to provide written consent to participate in the study.

Exclusion Criteria:

* Patients who have received BTX-A or BTX-B in the past in the skeletal muscle group under investigation or patients who have had an allergic response to BTX-A or BTX-B in the past.
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, or Amyotrophic Lateral Sclerosis. Females who are pregnant or breastfeeding. Subjects taking Aminoglycosides or other agents interfering with neuromuscular function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Volume and Cross-Sectional Area of Muscle | 36 Weeks
  The present pilot study is designed to assess the extent to which BTX-A (BOTOX) and BTX-B (MYOBLOC) cause muscle atrophy in spastic patients. The primary objective is to assess whether there is statistically significant difference in muscle atrophy between the two groups over a one-year period. Patient will complete a MRI of the tested muscle at baseline and at the end of the study. The MRI will be completed and read by the same radiologist throughout the study to account for inter rater variability. Note: The radiologist will be blinded to study treatment.

SECONDARY OUTCOMES:
Modified Ashworth Scale | 36 Weeks
  The secondary endpoint is improvement in spasticity using the Modified Ashworth Scale. We will review all measures with our statistician. Modified Ashworth scoring will be completed at every visit to evaluate the extent of spasticity before, during and after treatment of which will be conducted by the same rater throughout course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Pagan, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States